CLINICAL TRIAL: NCT02359019
Title: Phase II Study of MK-3475 as Maintenance Therapy in Extensive Stage Small Cell Lung Cancer (SCLC) Patients
Brief Title: MK-3475 as Maintenance Therapy in Extensive Stage SCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ammar Sukari, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-111; NCI-2015-00107 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-111 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Extensive Stage Small Cell Lung Carcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with extensive stage small cell lung cancer after completion of combination chemotherapy. Pembrolizumab may be effective in controlling small cell lung cancer for a longer period of time in patients with responsive or stable disease after completion of combination chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 defined progression-free survival (PFS) in extensive stage small cell lung cancer (SCLC) patients, who have complete response (CR), partial response (PR) or stable disease following minimum of 4 cycles of platinum (cisplatin or carboplatin) and etoposide.

SECONDARY OBJECTIVES:

I. To assess modified PFS in all patients enrolled. II. To assess overall survival of patients enrolled on the trial. III. To assess programmed cell death 1 ligand 1 (PD-L1) expression in archival tumor tissues and in circulating tumor cells (CTCs) and correlate the expression to RECIST defined PFS.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with extensive stage SCLC who have completed at least 4 cycles of platinum (carboplatin/cisplatin) and etoposide chemotherapy as their first line therapy and have responding or stable disease to this therapy are eligible for this study; patients who received platinum/etoposide previously for SCLC and it was repeated for recurrence will not be eligible
* Patients should be willing and able to provide written informed consent for the trial
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Demonstrate adequate organ function, all screening laboratories (labs) should be performed within 14 days of treatment initiation
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated* creatinine clearance >= 45 mL/min for subject with creatinine levels > 1.5 X institutional ULN; glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance [CrCl])

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 X ULN OR directed bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 1 week prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy greater than 10 mg/day or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or definitive radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent; patients who received palliative radiation to any site or prophylactic cranial radiation (=< 30 Gray [Gy]) or thoracic RT can start therapy with the study drug 7 days after the last day of radiation therapy as long as they have recovered from any adverse effects (i.e., =< grade 1 or at baseline) of such radiation therapy

  * Note: subjects with =< grade 2 neuropathy or adverse events that are not considered clinically meaningful such as alopecia are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; patient will be eligible if other malignancy is controlled and the treating physician determines that the patient's outcome is unlikely to be affected by the other tumor
* Has symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are clinically stable and any neurologic symptoms have returned to baseline, have no clinical evidence of new or enlarging brain metastases, and are not using steroids greater than prednisone 10mg/day or equivalent dose of another steroid" prior to start of trial treatment
* Has an active autoimmune disease, including a paraneoplastic syndrome of autoimmune nature, requiring systemic treatment other than chemotherapy for SCLC, within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires or required systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study
* Has evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-programmed cell death-1 (PD-1), anti-PD-L1, anti-PD-L2, anti-cluster of differentiation (CD)137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-02; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ammar Sukari, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (5):
- United States (5):
  - Rush University Medical Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 25
Age, Continuous [Median (Full Range); unit: years] | 65.6 [50.5 to 85.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 6
  Caucasian | 37
  Middle Eastern | 1
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: PFS Using RECIST 1.1
Description: Progression is defined using RECIST 1.1. PFS will be estimated with the standard Kaplan-Meier method, from which summary statistics of interest (median, 1-year rate, etc.) will be derived. Both point and 95% confidence interval estimates of PFS will be calculated.
Time Frame: Time from registration to time of progression, assessed up to 6 months after completion of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 45
months | 1.4 [1.3 to 2.8]

2. Secondary Outcome: Modified PFS Defined by RECIST as Progression That is Confirmed by a Second Scan at Least 4 Weeks Apart
Description: Progression is defined using RECIST 1.1. Estimated using standard Kaplan-Meier methods, from which the median and a 90% confidence interval will be calculated.
Time Frame: Time from registration to time of progression, assessed up to 6 months after completion of study treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 45
months | 6.3 [2.6 to 9.5]

3. Secondary Outcome: Overall Survival
Description: Estimated using standard Kaplan-Meier methods, from which the median and a 95% confidence interval will be calculated.
Time Frame: Time from registration to time of death, assessed up to 12 months after completion of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 45
months | 9.6 [7.0 to 12.0]

ADVERSE EVENTS:
Time Frame: Time from registration until off study, assessed up to 6 months after completion of study treatment.
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 34/45
Serious Adverse Events (participants affected / at risk) | 18/45
Other Adverse Events (participants affected / at risk) | 42/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=45)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Aspartate aminotransferase increase (Blood and lymphatic system disorders) | 2 (2)
Atrioventricular block complete (Vascular disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Cataract (Eye disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Endocrine disorders - Type 1 Diabetes (Endocrine disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6)
Lung infection- Pneumonia (Infections and infestations) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Neoplasms benign, malignant and (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pain (General disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Right lower/middle lobe pneumonia (Infections and infestations) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=45)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Alanine aminotransferase increased (Investigations) | 4 (5)
Alkaline phosphatase increased (Investigations) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Anxiety (Psychiatric disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9)
Constipation (Gastrointestinal disorders) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Creatinine increased (Investigations) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Dizziness (Nervous system disorders) | 9 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Edema limbs (General disorders) | 4 (4)
Fatigue (General disorders) | 18 (22)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (6)
Headache (Nervous system disorders) | 6 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 4 (10)
Hypothyroidism (Endocrine disorders) | 4 (5)
Lymphocyte count decreased (Investigations) | 5 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 12 (15)
Non-cardiac chest pain (General disorders) | 6 (8)
Pain (General disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6)
Platelet count decreased (Investigations) | 4 (6)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (23)
Rash acneiform (Skin and subcutaneous tissue disorders) | 8 (16)
Vomiting (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT02359019/Prot_SAP_000.pdf